CLINICAL TRIAL: NCT03727802
Title: TRK-250 - A Phase I, Double-Blind, Placebo-Controlled, Single and Multiple Inhaled Dose, Safety, Tolerability, and Pharmacokinetic Study of TRK-250 in Subjects With Idiopathic Pulmonary Fibrosis
Brief Title: Safety, Tolerability, and Pharmacokinetic Study of TRK-250 for Patients With Idiopathic Pulmonary Fibrosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Toray Industries, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 250IPF01
Record Dates: First submitted 2018-10-24; First posted 2018-11-01 (Actual); Results first posted 2023-10-23 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2022-06

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: TRK-250; Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TRK-250 (Experimental)
  Interventions: Drug: TRK-250
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TRK-250 — single and multiple doses (4 weeks)
  Arms: TRK-250
Drug: Placebo — single and multiple doses (4 weeks)
  Arms: Placebo

SUMMARY:
TRK-250 is a nucleic acid medicine that inhibits the progression of pulmonary fibrosis by selectively suppressing the expression of transforming growth factor-beta 1 (TGF-β1) protein, at the gene expression level. This study is a double-blind, randomized, placebo-controlled Phase I study. The primary objective of the study is to assess the safety and tolerability of single and multiple inhaled doses of TRK-250 in subjects with idiopathic pulmonary fibrosis (IPF).

ELIGIBILITY:
Inclusion Criteria:

* Clinical, radiographic, and histologic features consistent with the diagnosis of IPF
* SpO2 ≥90% at rest by pulse oximetry while breathing ambient air.
* FVC ≥50% of predicted.
* FEV1 ≥50% of predicted.
* Ratio of FEV1 to FVC ≥0.7.
* DLCO corrected for hemoglobin 30% to 79% of predicted, inclusive.

Exclusion Criteria:

* History of acute exacerbation of IPF or respiratory tract infection within 3 months prior to Screening.
* Planned surgery during the study.
* History of malignant tumor within 5 years prior to Screening.
* History of emphysema or clinically significant respiratory diseases (other than IPF).
* Other known causes of interstitial lung disease (eg, drug toxicities, environmental exposures, connective tissue diseases).
* End-stage fibrotic disease expected to require organ transplantation within 6 months.
* Taking a systemic corticosteroid, cytotoxic therapy, vasodilator therapy for pulmonary hypertension, or unapproved treatment for IPF within 4 weeks prior to Screening. (Treatment with pirfenidone or nintedanib, though not both concurrently, is permitted, provided that the subject has been on a stable dose for at least 4 weeks prior to Screening and it is anticipated the dose will remain unchanged throughout enrollment.)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2018-11-28 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Pulmonary Associates, Phoenix, Arizona
  - Cedars-Sinai Medical Center (CSMC) - Women's Guild Lung Institute, Los Angeles, California
  - UC Davis Medical Center, Sacramento, California
  - Advanced Pulmonary & Sleep Research Institute of Florida, Daytona Beach, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Pulmonary Disease Specialists, PA, d/b/a PDS Research. Kissimmee, FL, Kissimmee, Florida
  - Weill Cornell Medicine, New York, New York
  - PulmonIx LLC, Greensboro, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Medical University of South Carolina - Pulmonary & Critical Care Clinical Research Program, Charleston, South Carolina
  - The University of Texas Southwestern Medical Center, Dallas, Texas

REFERENCES:
- [Derived] Doi H, Atsumi J, Baratz D, Miyamoto Y. A Phase I Study of TRK-250, a Novel siRNA-Based Oligonucleotide, in Patients with Idiopathic Pulmonary Fibrosis. J Aerosol Med Pulm Drug Deliv. 2023 Dec;36(6):300-308. doi: 10.1089/jamp.2023.0014. Epub 2023 Sep 22. PMID 37738329

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 34 subjects were randomized to treatment, with 16 subjects in Part A and 18 subjects in Part B.
Groups:
- PartA:TRK-250 2mg; PartA:TRK-250 10mg; PartA:TRK-250 30mg; PartA:TRK-250 60mg: single dose of TRK-250
- PartA:Pooled Placebo: single dose of Placebo
- PartB:TRK-250 10mg; PartB:TRK-250 30mg; PartB:TRK-250 60mg: multiple doses (4 weeks) of TRK-250
- PartB:Pooled Placebo: multiple doses (4 weeks) of Placebo
Period: Overall Study
Arm/Group | PartA:TRK-250 2mg | PartA:TRK-250 10mg | PartA:TRK-250 30mg | PartA:TRK-250 60mg | PartA:Pooled Placebo | PartB:TRK-250 10mg | PartB:TRK-250 30mg | PartB:TRK-250 60mg | PartB:Pooled Placebo
Started | 3 | 3 | 3 | 3 | 4 | 4 | 4 | 4 | 6
Completed | 3 | 3 | 3 | 3 | 4 | 4 | 4 | 3 | 5
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PartA:TRK-250 2mg | PartA:TRK-250 10mg | PartA:TRK-250 30mg | PartA:TRK-250 60mg | PartA:Pooled Placebo | PartB:TRK-250 10mg | PartB:TRK-250 30mg | PartB:TRK-250 60mg | PartB:Pooled Placebo | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 4 | 4 | 4 | 6 | 34
Age, Customized [Mean (Full Range); unit: years]
  Age | 74 [70 to 76] | 70 [66 to 73] | 76 [70 to 80] | 69 [66 to 74] | 75 [67 to 79] | 64 [48 to 74] | 70 [59 to 75] | 74 [66 to 78] | 75 [70 to 77] | 72 [48 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 7
  Male | 1 | 2 | 2 | 2 | 4 | 4 | 4 | 2 | 6 | 27
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 3 | 3 | 2 | 3 | 4 | 4 | 4 | 4 | 6 | 33
  Race: Black or African Black or African American | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Adverse Events
Description: Number of patients reporting Adverse Events Number of patients by severity reporting Adverse Events
Time Frame: Up to 14 days after last dose
Measure: Count of Participants; unit: Participants
Arm/Group | PartA:TRK-250 2mg | PartA:TRK-250 10mg | PartA:TRK-250 30mg | PartA:TRK-250 60mg | PartA:Pooled Placebo | PartB:TRK-250 10mg | PartB:TRK-250 30mg | PartB:TRK-250 60mg | PartB:Pooled Placebo
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 4 | 4 | 4 | 4 | 6
Participants
  Subjects with AEs | 1 | 0 | 3 | 2 | 1 | 3 | 2 | 3 | 3
  Mild(Severity) | 0 | 0 | 2 | 1 | 1 | 2 | 1 | 0 | 3
  Moderate(Severity) | 1 | 0 | 1 | 1 | 0 | 1 | 1 | 2 | 0
  Severe(Severity) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Up to 14 days after last dose
Arm/Group | PartA:TRK-250 2mg | PartA:TRK-250 10mg | PartA:TRK-250 30mg | PartA:TRK-250 60mg | PartA:Pooled Placebo | PartB:TRK-250 10mg | PartB:TRK-250 30mg | PartB:TRK-250 60mg | PartB:Pooled Placebo
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/4 | 0/4 | 0/4 | 0/4 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/3 | 0/4 | 0/4 | 0/4 | 1/4 | 0/6
Other Adverse Events (participants affected / at risk) | 1/3 | 0/3 | 3/3 | 2/3 | 1/4 | 3/4 | 2/4 | 3/4 | 3/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PartA:TRK-250 2mg (N=3) | PartA:TRK-250 10mg (N=3) | PartA:TRK-250 30mg (N=3) | PartA:TRK-250 60mg (N=3) | PartA:Pooled Placebo (N=4) | PartB:TRK-250 10mg (N=4) | PartB:TRK-250 30mg (N=4) | PartB:TRK-250 60mg (N=4) | PartB:Pooled Placebo (N=6)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PartA:TRK-250 2mg (N=3) | PartA:TRK-250 10mg (N=3) | PartA:TRK-250 30mg (N=3) | PartA:TRK-250 60mg (N=3) | PartA:Pooled Placebo (N=4) | PartB:TRK-250 10mg (N=4) | PartB:TRK-250 30mg (N=4) | PartB:TRK-250 60mg (N=4) | PartB:Pooled Placebo (N=6)
Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bundle branch block right (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Glaucoma (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eosinophil count increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Heart rate irregular (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/02/NCT03727802/Prot_000.pdf
  • Statistical Analysis Plan (2019-06-25): https://cdn.clinicaltrials.gov/large-docs/02/NCT03727802/SAP_001.pdf